CLINICAL TRIAL: NCT01686711
Title: A Phase 4, Multicenter, Randomized, Double-blind, Parallel-group, Comparative Study to Evaluate the Efficacy and Safety of AD-4833 When Orally Administered Once Daily as add-on to SYR-322 Versus SYR-322 Alone in the Treatment of Type 2 Diabetes Mellitus With Inadequate Glycemic Control Despite Treatment With SYR-322 in Addition to Diet and/or Exercise Therapy
Brief Title: A Double-blind, Parallel Group, Comparative Study of Coadministration AD-4833 and SYR-322
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: SYR-322-4833/CCT-901; U1111-1132-3209 (Registry Identifier: WHO); JapicCTI-121916 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2012-08-31; First posted 2012-09-18 (Estimated); Last update posted 2023-08-31 (Actual); Status verified 2023-08

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus | interventions — Pioglitazone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- SYR-322 25 mg , AD-4833 15 mg (Experimental)
  Interventions: Drug: AD-4833 15 mg
- SYR-322 25 mg , AD-4833 30 mg (Experimental)
  Interventions: Drug: AD-4833 30 mg
- SYR-322 25 mg , AD-4833 placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AD-4833 15 mg
  Arms: SYR-322 25 mg , AD-4833 15 mg
Drug: AD-4833 30 mg
  Arms: SYR-322 25 mg , AD-4833 30 mg
Drug: Placebo
  Arms: SYR-322 25 mg , AD-4833 placebo

SUMMARY:
To evaluate the efficacy and safety of coadministration AD-4833 and SYR-322 in patients with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria:

* Those judged to be capable of understanding and complying with protocol requirements by the investigator or subinvestigator.
* Those who can sign and date a written, informed consent form prior to the initiation of any study procedures.

Exclusion Criteria:

* Those with concurrent serious cardiac disease, serious cerebrovascular disorder, or serious pancreatic or hematological disease etc.
* Others who are assessed to be ineligible for the study by the investigator or subinvestigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 207 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Glycosylated Hemoglobin (HbA1c) | 16 weeks
  Measurement of change in HbA1c (ratio of hemoglobin bound to glucose)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda (Note: This product was divested to Teijin Pharma Limited in 2023)
Locations (25):
- Japan (25):
  - Hirosaki-shi, Aomori
  - Kisaratsu-shi, Chiba
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Kitakyushu-shi, Fukuoka
  - Kurume-shi, Fukuoka
  - Fukuyama-shi, Hiroshima
  - Hiroshima, Hiroshima
  - Sapporo, Hokkaido
  - Koga-shi, Ibaraki
  - Yokohama, Kanagawa
  - Kumamoto, Kumamoto
  - Miyazaki, Miyazaki
  - Suita-shi, Osaka
  - Koshigaya-shi, Saitama
  - Ōtsu, Shiga
  - Chiyoda-ku, Tokyo
  - Chuo-ku, Tokyo
  - Itabashi-ku, Tokyo
  - Meguro-ku, Tokyo
  - Minato-ku, Tokyo
  - Ohta-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Toyama, Toyama
  - Shimonoseki-shi, Yamaguchi